CLINICAL TRIAL: NCT06178224
Title: Determination of Quantitative Beta-hCG Levels in Patients Through Alternative and Less Invasive Sample Types
Brief Title: Determining Beta-hCG Levels in Patients Through Alternative Sample Types
Status: Completed | Type: Observational
Sponsor: Simple HealthKit (Industry)
Collaborators: Planned Parenthood Federation of America (Other); Planned Parenthood Great Northwest, Hawai'I, Alaska, Indiana, Kentucky (Unknown)
Responsible Party: Sponsor
Other Study IDs: SHK_007
Record Dates: First submitted 2023-11-29; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Pregnancy Related; Abortion
Keywords: Simple HealthKit

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples collected from each user are:
  Urine Saliva Serum dried blood spot (DBS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants (qualified): This arm consists of participants who are able to collect all sample types No intervention is administered

SUMMARY:
This study is to determine if there is any quantifiable correlation between serum beta hCG and dried blood spot (DBS) beta hCG levels. This data will be used to develop a less invasive collection method to determine quantitative hCG levels.

DETAILED DESCRIPTION:
A cohort of 40 individuals at various stages of pregnancy or medical abortion will be recruited for the study. Each participant will provide biospecimens that include the following: serum, saliva, urine, and dried blood spot (DBS). These samples will be collected and stored at the clinic under appropriate storage conditions until they can be shipped, under dry ice, to the testing lab. Once samples arrive at the lab, serum samples will be thawed and prepared to run on an ECL analyzer to determine reference beta hCG values in mIU/mL for each participant.

Samples will be run as they are received by the lab. The initial 10-12 samples will be used to evaluate study feasiblility and determine if there is one sample type that performs better than the others. The other matched sample types will be processed and run on the ECL analyzer. The values for beta hCG mIU/mL of the other sample types will then be compared to the matched serum to determine if there are any consistent correlations.

In the first 10-12 samples, if one sample type is shown to perform better than the others, the study will shift focus towards prioritizing the analysis of that particular sample type in regards to correlation with serum. If more than one sample type is shown to perform well, then those sample types will be equally prioritized. If no sample type shows any correlation, the study will end.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Have not taken antibiotics in the last 21 days
* Are here for services related to a current or recent pregnancy
* Agree to provide all required samples
* Have not previously participated in this study

Exclusion Criteria:

* Are under18 years old
* Have taken antibiotics in the last 21 days
* Are not here for services related to a current or recent pregnancy
* Disagree or unable to provide all required samples
* Have previously participated in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consists of individuals who are of 18 years or older that are currently pregnant or undergoing medical abortion. All of the participants will come from affiliated Planned Parenthood clinics.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Correlation of matched serum and DBS samples for detection of beta hCG levels using an ECL analyzer. | 2-24 hours
  It was determine that serum and DBS samples show a consistent correlation. DBS beta hCG levels can be converted to reflect those of serum beta hCG. By utilization of a dilution factor, DBS beta hCG levels matched that of serum beta hCG levels with an average accuracy of 94.8%.
  Serum samples were run on an analyzer to obtain reference values in mIU/mL. Dried blood spot (DBS) samples, that were matched for both time of collection and patient, were extracted with an elution buffer coupled with agitation. This eluate was run on the same analyzer as the serum samples and the resulting beta hCG levels in mIU/mL were corrected with a dilution factor and compared to the serum reference values.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Berry, MD, Principal Investigator — Planned Parenthood Great Northwest, Hawai'I, Alaska, Indiana, Kentucky
Locations (1):
- Planned Parenthood of the Great Northwest, Hawai'i, Alaska, Indiana and Kentucky, Tacoma, Washington, United States